CLINICAL TRIAL: NCT04966260
Title: Virtual Reality Therapy to Improve Physical and Psychological Symptoms and Quality of Life for End-of-life Patients on a Palliative Care Unit: a Randomized Controlled Study
Brief Title: Virtual Reality Therapy to Improve Physical and Psychological Symptoms and Quality of Life for End-of-life Patients on a Palliative Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baycrest (Other)
Responsible Party: Principal Investigator, Ginah Kim, Staff Physician Palliative Care Unit, Baycrest
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 21-15
Record Dates: First submitted 2021-06-29; First posted 2021-07-19 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: End-of-Life; Physical Suffering; Psychological Distress
Keywords: Palliative Care; Symptom management; Virtual Reality
MeSH Terms: conditions — Death; Pain

STUDY DESIGN:
Intervention Model Description: This is a small randomized controlled trial conducted in a study population of patients admitted to a geriatric palliative care unit. The clinical team will determine if the patient is eligible for the study. Patients and families/friends of patients who are randomized to the personalized VR will be consented over the telephone by the research assistant., Participants will then be randomly assigned into one of the three study arms: comparator, standardized VR or personalized VR, on a 1:1:1 basis using computer-generated random numbers and a block size of 3 without additional stratification.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standardized Virtual Reality (Experimental): Participants in the standard virtual reality (VR) group will choose from the general library of VR experiences. Participants will be asked to select an experience they desire but have never experienced in person. The session will be facilitated by the therapeutic recreation staff on the unit.
  Interventions: Other: Standardized Virtual Reality
- Personalized Virtual Reality (Experimental): There are two types of personalized VR: 1) Family/friends provide personalized content (e.g., life stories, photos, videos) that will be used during the VR session. Family/friends of participants in the personalized VR group will have the opportunity to upload custom photos, videos, life stories or capture their own 360° footage of family events using a GoPro camera that will be loaned to them for the study. This content will be uploaded to a cloud-based portal. 2) If the family/friends of those in the personalized VR arm are unavailable/unable/unwilling to provide personalized content the participant will select a video from the VR library of an experience that is personally memorable to them, such as their childhood hometown, a favourite vacation destination. The session will be facilitated by the therapeutic recreation staff on the unit.
  Interventions: Other: Personalized Virtual Reality
- Two-Dimensional Video (Active Comparator): Participants in the active comparator group will choose a two-dimensional video such as a mountain view, ocean view or safari. Participants will view the two-dimensional video on an iPad and the session will be facilitated by the therapeutic recreation staff on the unit.
  Interventions: Other: Control

INTERVENTIONS:
Other: Standardized Virtual Reality — This is a one session intervention, where participants will be asked to wear a VR headset and view a three-dimensional standard VR video. The activity session will be approximately 15 minutes in length. Prior to starting the intervention, the therapeutic recreation staff will explain the activity and familiarize participants with the VR headset.
  Arms: Standardized Virtual Reality
Other: Control — This is a one session intervention, where participants will be asked to view a two-dimensional video on an iPad. The activity session will be approximately 15 minutes in length. Prior to starting the activity session, the therapeutic recreation staff will explain the activity.
  Arms: Two-Dimensional Video
Other: Personalized Virtual Reality — This is a one session intervention, where participants will be asked to wear a VR headset and view a three-dimensional personalized VR video. The activity session will be approximately 15 minutes in length. Prior to starting the intervention, the therapeutic recreation staff will explain the activity and familiarize participants with the VR headset.
  Arms: Personalized Virtual Reality

SUMMARY:
People with advanced and life-threatening illnesses experience challenges across multiple domains of function including physical, psychological, social, and spiritual. The benefits of non-pharmacological interventions for palliative care patients are well recognized, but are relatively under-utilized. Virtual Reality (VR) therapy may help address these challenges and be a valuable addition to the current therapies used in palliative care.

VR is a computer generated, three-dimensional environment that individuals can explore and interact with using specialized equipment such as a head-mounted display with internal sensors. VR has been increasingly adapted for applications in healthcare, as a simulation for medical training and an intervention tool to impact pain management, stress and anxiety. VR has the potential to improve both physical and psychological symptoms in patients with terminal illnesses.

The current study is a small randomized controlled trial to understand the impact of VR on physical symptoms, psychological symptoms and quality of life in patients at the end of life. Participants will be randomized to a single comparator session, single session of standard VR, or single session of personalized VR. The comparator arm will consist of participants viewing an ordinary two-dimensional video on an iPad such as a peaceful nature scene. The standard VR arm will consist of participants viewing a "bucket list" experience self-selected from a VR library i.e. an experience the participant desires but has never experienced. The personalized VR arm will consist of participants viewing content that is personally meaningful to them. This content will be obtained through either a) family/friends creating a personalized video (e.g. video footage of their summer cottage) or b) the participant will select an experience from the VR library that is personally meaningful (e.g. visiting their honeymoon destination, exploring their childhood hometown, etc.) if option a) is not possible.

Participants will complete self-report questionnaires about their physical and psychological symptoms and quality of life before and after the intervention (two days and seven days post intervention). Participants will also complete a feedback survey to evaluate their satisfaction with the intervention. Surveys will be administered by the research assistant.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to Baycrest PCU
* Capable to consent to the study
* Able to complete the outcome measures through a telephone interview with a research assistant
* Estimated prognosis ≥3 weeks
* At least 2 or more ESAS scores of 4 or greater within the week of the intervention
* English speaking

Exclusion Criteria:

* Intractable nausea/vomiting
* History of seizures or epilepsy
* Vision and/or hearing impairment that cannot be accommodated e.g. pocket talker
* Any abnormalities of the head preventing use of the headset
* Patients who are too unwell to participate based on the opinion of the clinical team

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
Change in Edmonton Symptom Assessment Scale (ESAS) Score | Pre-intervention, post-intervention (same day immediately after intervention), 2 day follow up, 7 day follow up
  The ESAS is a self-report measure used to assist in the assessment of pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, wellbeing, and shortness of breath (Bruera, Kuehn, Miller, Selmser, & Macmillan, 1991). The severity of the symptom at the time of the assessment is rated from zero to ten, with zero meaning the symptom is absent and ten meaning worst possible severity. For the purpose of the study the ESAS was modified to include two additional items, headache and dizziness.
  Analysis of the ESAS scores across the different time points will help determine whether VR effects are transient (within 24 hours) or sustained (after 2 and 7 days).
Change in Missoula-VITAS Quality of Life Index (MVQOLI) | Pre-intervention, post-intervention (same day immediately after intervention), 2 day follow up, 7 day follow up
  The MVQOLI evaluates subjective quality of life among people living with advanced, life-threatening illness by assessing the domains of symptoms, function, interpersonal, wellbeing, and transcendence (Schwartz, Merriman, Reed, & Byock, 2005). Each domain includes three Likert-scale evaluation questions.
  Analysis of the MVQOLI scores across the different time points will help determine whether VR effects are transient (within 24 hours) or sustained (after 2 and 7 days).

CONTACTS AND LOCATIONS:
Overall Officials: Ginah Kim, MD, Principal Investigator — Baycrest
Locations (1):
- Baycrest Health Sciences, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson F, Downing GM, Hill J, Casorso L, Lerch N. Palliative performance scale (PPS): a new tool. J Palliat Care. 1996 Spring;12(1):5-11. PMID 8857241
- [Background] Hui D, Shamieh O, Paiva CE, Perez-Cruz PE, Kwon JH, Muckaden MA, Park M, Yennu S, Kang JH, Bruera E. Minimal clinically important differences in the Edmonton Symptom Assessment Scale in cancer patients: A prospective, multicenter study. Cancer. 2015 Sep 1;121(17):3027-35. doi: 10.1002/cncr.29437. Epub 2015 Jun 8. PMID 26059846
- [Background] Schwartz CE, Merriman MP, Reed G, Byock I. Evaluation of the Missoula-VITAS Quality of Life Index--revised: research tool or clinical tool? J Palliat Med. 2005 Feb;8(1):121-35. doi: 10.1089/jpm.2005.8.121. PMID 15662181